CLINICAL TRIAL: NCT02478281
Title: A One-Period, Single-Dose, Safety, Tolerability, and Pharmacokinetic Study of Methylene Blue Injection United States Pharmacopeia (USP) Following a 1 mg/kg Intravenous Dose in Healthy Adult Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetic Study of Methylene Blue Following a 1 mg/kg Intravenous Dose in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1MBL12002
Record Dates: First submitted 2015-04-28; First posted 2015-06-23 (Estimated); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2018-01

CONDITIONS: Methemoglobinemia; Congenital Methemoglobinemia
MeSH Terms: conditions — Methemoglobinemia; Congenital Methemoglobinemia | interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methylene Blue Injection, United States Pharmacopeia (USP) (Experimental): Single dose of Methylene Blue Injection, USP at a dose of 1 mg/kg solution per kg given intravenously over a period of approximately 5 minutes.
  Interventions: Drug: Methylene Blue

INTERVENTIONS:
Drug: Methylene Blue

SUMMARY:
A Phase 1 trial to assess the single-dose safety, tolerability, and pharmacokinetic (PK) of Methylene Blue Injection, USP 1 mg/kg in healthy adult volunteers.

DETAILED DESCRIPTION:
This is an open-label, single-center, one-arm, safety, tolerability, and PK study in healthy male and female volunteers of Methylene Blue Injection, USP. Following an overnight fast, twelve healthy adult male and female volunteers will receive a single dose of study drug at a dose of 1 mg/kg solution per kg given intravenously over a period of 5 minutes followed by serial venous blood sampling at 0.042, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 16, 36, 48, and 72 hours postdose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female volunteers, 18-60 years of age, inclusive.
* Weigh at least 52 kg for males and 45 kg for females and within the normal range according to accepted normal values of the Body Mass Index (BMI) chart 18.5-29.9 kg/m² inclusive.
* Medically healthy with no clinically significant laboratory profiles, vital signs, or ECG's; as deemed by the PI.
* For females of childbearing potential: either be sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or be using acceptable birth control methods. Female subjects who claim to be sexually inactive, but become sexually active during the course of the study must agree to use a barrier method (e.g. condom, diaphragm)with spermicide from the time of the start of sexual activity through at least 30 days following dosing. In addition, female subjects of childbearing potential will be advised to remain sexually inactive or to keep the same birth control method for at least 30 days following dosing.
* Females of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to Day 1:

  * Hysteroscopic tubal ligation (with a copy of the confirmation test) and be using a barrier method (condom or diaphragm) and spermicide throughout the study;
  * Bilateral tubal ligation and be using a barrier method (condom or diaphragm) and spermicide throughout the study;
  * Hysterectomy;

    * Bilateral oophorectomy or be postmenopausal with amenorrhea for at least 1 year prior to Day 1 and follicle stimulating hormone (FSH) serum levels ≥ 40 milli-International Units per mL (mIU/mL). Females on hormone replacement therapy may be deemed eligible for participation in the study even if their FSH levels < 40 mIU/mL, if they are able to provide documentation of FSH levels 40 mIU/mL before initiation of hormone replacement therapy.
* Males must use condom with spermicide when engaged in sexual activity and must agree to refrain from sperm donation from check-in through 90 days postdose.
* Willing to answer inclusion and exclusion criteria questionnaire at check-in.
* Give voluntary written informed consent to participate in the study.
* Be able to comply with the protocol and the assessments therein.

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease in the opinion of the PI.
* History or presence of alcoholism within the past 2 years.
* History or presence of drug abuse within the past 2 years.
* History or presence of hypersensitivity or idiosyncratic reaction to Methylene Blue.
* History or presence of Glucose-6-Phosphate Dehydrogenase (G6PD) dehydrogenase deficiency, retinopathy, blood disorder, myasthenia gravis, psoriasis, epilepsy, clinically significant allergies (except for mild forms of hay fever), or any other clinically significant medical condition, which in the opinion of the PI, might interfere with study participation.
* History or laboratory evidence of renal insufficiency.
* Any screening laboratory test with clinically significant abnormalities in the opinion of the PI (including cell blood count, creatinine, or liver function tests).
* Have used any drug that acts as a serotonin reuptake inhibitor (SRIs) e.g. selective serotonin reuptake inhibitors (SSRIs), tricyclic antidepressants (TCAs), norepinephrine-dopamine reuptake inhibitors (NDRIs), triptans, or ergot alkaloids within 30 days (or 5 half-lives of the compound, whichever is longer) prior to study drug dosing.
* Female subjects who are pregnant or lactating, or female subjects who are likely to become pregnant during the study.
* Had positive results for the urine drug/alcohol screen at screening or check-in.
* Had positive results at screening for HIV, HBsAg, or hepatitis C virus (HCV).
* Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
* Heart rate is lower than 40 bpm or higher than 99 bpm at screening.
* QTc interval is >430 msec (males) or >450 msec (females) or deemed clinically abnormal by the PI or use of any drug or agent suspected of causing QT prolongation or torsade de pointes within 14 days (or 5 half- lives of the compound, whichever is longer) prior to study drug dosing.
* Have been on a special diet (for whatever reason) within the 28 days prior to study drug dosing, and throughout the study.
* Have made a donation of blood or had significant blood loss within 56 days prior to study drug dosing.
* Have made a plasma donation within 7 days prior to study drug dosing.
* Have received Methylene Blue within 72 hours prior to study drug dosing.
* Have participated in another clinical trial within 30 days (or 5 half-lives of the compound, whichever is longer) prior to study drug dosing.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fareeda Hosein, MD, Principal Investigator — Celerion

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 1 investigator center.
Pre-assignment Details: Of the 12 participants enrolled, all met eligibility requirements and were treated.
Groups:
- Methylene Blue Injection, USP: Single dose of Methylene Blue Injection, United States Pharmacopeia (USP) at a dose of 1 mg/kg solution per kg given intravenously over a period of approximately 5 minutes.
  Methylene Blue
Period: Overall Study
Arm/Group | Methylene Blue Injection, USP
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat
Groups:
- Methylene Blue Injection, USP: Single dose of Methylene Blue Injection, USP at a dose of 1 mg/kg solution per kg given intravenously over a period of approximately 5 minutes.
  Methylene Blue
Arm/Group | Methylene Blue Injection, USP
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Weight [Mean (Standard Deviation); unit: kilograms] | 76.13 (11.75)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) From Time Zero to the Time of Last Quantifiable Concentration (AUC 0-t)
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample; AUC 0-t is defined as AUC from time 0 to the last data point
Time Frame: pre-dose, 0.042, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 16, 36, 48, and 72 hours post-dose
Population: Intent to treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Methylene Blue Injection, USP
Number analyzed (Participants) | 12
ng*hr/mL | 2600.09 (28.7)

2. Primary Outcome: Area Under the Curve From Time Zero Extrapolated to Infinity (AUC 0-∞)
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC 0-∞ is defined as area under the concentration vs. time curve from zero to infinity.
Time Frame: pre-dose, 0.042, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 16, 36, 48, and 72 hours post-dose
Population: Intent to treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Methylene Blue Injection, USP
Number analyzed (Participants) | 12
ng*hr/mL | 2967.09 (27.9)

3. Primary Outcome: The Percent of Extrapolated Area Under the Curve (AUC%Extrap)
Description: The AUC%extrap refers to the fraction of the total AUC that is due to the extrapolated AUC
Time Frame: pre-dose, 0.042, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 16, 36, 48, and 72 hours post-dose
Population: Intent to treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent of AUC
Arm/Group | Methylene Blue Injection, USP
Number analyzed (Participants) | 12
Percent of AUC | 11.72 (32.9)

4. Primary Outcome: Area Under the Curve Ratio (AUCR)
Description: AUCR refers to the ratio of AUC 0-t to AUC 0-∞.
Time Frame: pre-dose, 0.042, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 16, 36, 48, and 72 hours post-dose
Population: Intent to treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent
Arm/Group | Methylene Blue Injection, USP
Number analyzed (Participants) | 12
Percent | 87.63 (4.6)

5. Primary Outcome: Total Body Clearance (CL)
Description: CL refers to the Dose/AUC 0-∞
Time Frame: pre-dose, 0.042, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 16, 36, 48, and 72 hours post-dose
Population: Intent to treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Methylene Blue Injection, USP
Number analyzed (Participants) | 12
L/hour | 19.02 (22.5)

6. Primary Outcome: Maximum Measured Plasma Concentration (Cmax)
Description: Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: pre-dose, 0.042, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 16, 36, 48, and 72 hours post-dose
Population: Intent to Treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Methylene Blue Injection, USP
Number analyzed (Participants) | 12
ng/mL | 457.34 (41.9)

7. Primary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Tmax refers to the time it takes for a drug to reach maximum concentration
Time Frame: pre-dose, 0.042, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 16, 36, 48, and 72 hours post-dose
Population: Intent to Treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Methylene Blue Injection, USP
Number analyzed (Participants) | 12
Hours | 0.217 (126.7)

8. Primary Outcome: Terminal Elimination Half-life (T1/2)
Description: T1/2 refers to the time taken for concentration of a drug to decrease from its maximum concentration to half of Cmax
Time Frame: pre-dose, 0.042, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 16, 36, 48, and 72 hours post-dose
Population: Intent to Treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Methylene Blue Injection, USP
Number analyzed (Participants) | 12
Hours | 15.908 (46.3)

9. Primary Outcome: Terminal Elimination Rate Constant (Lambda Z)
Description: Lambda Z refers to the terminal elimination phase for drug plasma concentration vs. time data
Time Frame: pre-dose, 0.042, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 16, 36, 48, and 72 hours post-dose
Population: Intent to Treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Methylene Blue Injection, USP
Number analyzed (Participants) | 12
1/hour | 0.04357 (46.3)

10. Primary Outcome: Volume of Distribution (Vz) Based on Terminal Phase
Description: Vz refers to the ratio of amount of drug in a body (dose) to concentration of the drug that is measured in blood, plasma, and un-bound in interstitial fluid.
Time Frame: pre-dose, 0.042, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 16, 36, 48, and 72 hours post-dose
Population: Intent to treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Groups:
- Methylene Blue Injection, United States Pharmacopeia (USP): Single dose of Methylene Blue Injection, USP at a dose of 1 mg/kg solution per kg given intravenously over a period of approximately 5 minutes.
  Methylene Blue
Arm/Group | Methylene Blue Injection, United States Pharmacopeia (USP)
Number analyzed (Participants) | 12
Liters | 436.557 (40.3)

11. Primary Outcome: Mean Residence Time (MRT)
Description: MRT refers to the average amount of time that a drug molecule spends in the body before being removed
Time Frame: pre-dose, 0.042, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 16, 36, 48, and 72 hours post-dose
Population: Intent to treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Methylene Blue Injection, USP
Number analyzed (Participants) | 12
Hours | 17.677 (39.8)

ADVERSE EVENTS:
Time Frame: 4 days
Description: An adverse event was defined as any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research
Arm/Group | Methylene Blue Injection, USP
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 10/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylene Blue Injection, USP (N=12)
Tachycardia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Infusion site pain (General disorders) | 5 (5)
Infusion site pruritus (General disorders) | 1 (1)
Vessel puncture site hematoma (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No